CLINICAL TRIAL: NCT04266054
Title: Stories for Change: Digital Storytelling for Diabetes Self-Management Among Somali Adults
Acronym: S4C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jane W. Njeru, M.B., Ch.B., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 19-008588
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will view the 12-minute digital storytelling intervention that has been previously pilot-tested, in addition to usual clinical care
  Interventions: Behavioral: Digital Storytelling Intervention
- Control (No Intervention): The comparison group will receive usual clinical care.

INTERVENTIONS:
Behavioral: Digital Storytelling Intervention — 12-minute digital storytelling intervention in Spanish, with four individuals explaining their personal Type 2 Diabetes stories.
  Arms: Intervention

SUMMARY:
Somali adults are more likely to have type 2 diabetes mellitus (T2D) and more likely to die from the disease than non-Somali whites. These disparities are mediated, in part, by less healthful levels of physical activity, dietary quality, medication adherence, and self-monitoring of blood glucose than non-Somali whites. Innovative approaches that arise from affected communities are needed to address these health disparities.

Community-based participatory research (CBPR) has been successful in targeting health issues among Somali and immigrant populations; CBPR is an effective approach for addressing health behaviors in a sociocultural context. In 2004, the research team developed a CBPR partnership between immigrant communities and academic institutions called Rochester Healthy Community Partnership (RHCP)

Storytelling or narrative-based interventions are designed to incorporate culture-centric health messaging to promote behavior change among vulnerable populations. Digital storytelling interventions are narrative-based videos elicited through a CBPR approach to surface the authentic voices of individuals overcoming obstacles toward engaging in health promoting behaviors to shape positive health behaviors of viewers through influences on attitudes and beliefs.

RHCP partners from Somali communities identified T2D as a priority area for intervention, and have co-created each of the formative phases leading up to this proposal. Narrative theory and social cognitive theory formed the conceptual basis for intervention development. The study team conducted surveys and focus groups to derive the approach and personnel for building an authentic intervention that was created in a digital storytelling workshop where stories about diabetes self-management were captured, recorded, and edited to derive the final intervention products in video format. The respective digital storytelling videos will be pilot tested with 80 patients in Rochester, MN. In a mirror project for Hispanic adults, the intervention was rated as highly acceptable, culturally relevant, and perceived as efficacious for motivating behavioral change.

The overall objective of this project is therefore to assess the efficacy of a digital storytelling intervention derived through a CBPR approach on self-management of T2D among Somali adults.

DETAILED DESCRIPTION:
The study team will conduct a two-group randomized controlled trial in a primary care clinical setting at Mayo Clinic in Rochester, MN with Somali adults with poorly controlled T2D (hemoglobin A1c≥8%). The intervention group will view the 12-minute digital storytelling video. Both the intervention and comparison groups will receive diabetes education and resource cards, as well as usual clinical care. The primary outcome will be glycemic control as measured by hemoglobin A1c 3 months after intervention delivery. Secondary outcomes will include diabetes self-management behaviors, blood pressure, LDL-cholesterol, and body mass index. The impact of concomitant covariates, including sex, age, and socio-economic status, on the sensitivity of the intervention effect will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identifies as Somali
2. Between 18 and 70 years of age.
3. Receives primary care at Mayo Clinic ECH.
4. Visited the primary care site at least once in the least twelve months.
5. Intention to continue receiving care at the clinic for the next six months.
6. Diagnosis of T2D in medical record.
7. T2D diagnosis for six months or longer.
8. Most recent hemoglobin A1c≥8%.

Exclusion Criteria:

1. Not eligible if someone in the same household is participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control as measured by hemoglobin A1c. Hemoglobin A1c will be measured from whole blood samples obtained and analyzed in a blinded fashion. | 6 months
  The rationale for use of hemoglobin A1c as an indicator of diabetes control is based on national and regional data that demonstrate significant disparities in reaching hemoglobin A1c targets for Somali populations compared with non-Somali whites. The importance of glycemic control as part of the comprehensive management of diabetes is well documented, and hemoglobin A1c testing is a well-established strategy to monitor glycemic control in patients with diabetes.

SECONDARY OUTCOMES:
Diabetes self-management behaviors will be assessed with the Summary of Diabetes Self-Care Activities Measure (SDSCA). | 6 months
  This is a brief survey instrument to assess the following domains: general diet, specific (diabetes) diet, physical activity, diabetes medication use, and blood glucose monitoring. In a 2009 review of psychometric tools to assess diabetes self-management behaviors, the SDSCA was one of only three instruments to meet all appraisal criteria113. The SDSCA is also the most commonly used instrument for these domains worldwide, with good validity evidence in several languages. The SDSCA will be administered by the same language-congruent study staff at each measure.
Seated blood pressure measurements (systolic and diastolic) will be made on the right arm using an automated blood pressure device after sitting quietly for five minutes. | 6 months
  Blood pressure will be measured three times; the average of the second and third readings will be used in statistical analyses.
Body mass index | 6 months
  Weight will be measured to the nearest 0.1 kg using a clinical scale. Height will be measured in cm with a stadiometer. BMI is calculated as weight (kg)/height squared (m2).
Total cholesterol, HDL cholesterol, will be measured from the same blood sample used to derive the outcome measure. LDL-cholesterol will be calculated for each participant based on these values. | 3 months
  Baseline LDL-cholesterol values will be drawn at the baseline study visit. Cholesterol values at 3 months will be drawn at the 3 month study visit. Subsequent cholesterol levels will not be drawn or abstracted.
triglycerides will be measured from the same blood sample used to derive the outcome measure. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jane Njeru, MB, ChB, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials